CLINICAL TRIAL: NCT01384630
Title: A Phase II Open Label Study of the Safety, Pharmacokinetics, and Efficacy of a True Human Anti-inflammatory Therapeutic Antibody (RA-18C3) in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: Safety, Pharmacokinetics, and Efficacy of RA-18C3 in Subjects With Moderate to Severe Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-PT019
Record Dates: First submitted 2011-06-08; First posted 2011-06-29 (Estimated); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — bermekimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single group (Other)
  Interventions: Drug: RA-18C3

INTERVENTIONS:
Drug: RA-18C3 — 200 mg subcutaneous injection

SUMMARY:
This is a 73-day phase II, open label trial of the true human monoclonal antibody RA-18C3 in subjects with moderate to severe plaque psoriasis. Ten (10) subjects will receive 200 mg of RA-18C3 via subcutaneous injection. Subjects will receive injections at Days 0, 21, and 42 for a total of 3 injections. Study drug will be administered under close observation in a facility equipped to handle medical emergencies. Subjects will not be discharged from the facility until at least 1 hour following the end of the injection or 1 hour after their vital signs have stabilized. Safety will be assessed by pre- and post-treatment serial measurements of vital signs, clinical laboratory assessments, and the recording of adverse clinical events.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 18 years of age or older
2. Diagnosis of plaque psoriasis for ≥ 6 months; INCLUDING subjects with chronic guttate lesions.
3. Psoriasis area-and-severity index (PASI) score of ≥ 12
4. Involvement of ≥ 5% of body-surface area
5. For female subjects of childbearing age, a negative urine pregnancy test at screening and at specified time points throughout the trial. For subjects with reproductive potential, a willingness to utilize adequate, double barrier contraception during the study and including 3 months after study completion. Sexually active men must use an accepted method of contraception during the study and including 3 months after study completion.
6. Signed and dated Institutional Review Board (IRB) approved informed consent before any protocol-specific screening procedures are performed

Exclusion Criteria:

1. Treatment with any biologicals or investigational agents within the last 4 weeks (or 5 half-lives, whichever is longer).
2. Treatment with conventional systemic psoriasis therapy within last 4 weeks
3. Treatment with phototherapy within the last 4 weeks
4. Topical psoriasis treatment with the last 2 weeks
5. History of uncontrolled diabetes, unstable ischemic heart disease, active inflammatory bowel disease, active peptic ulcer disease, recent stroke (within 3 months), ongoing congestive heart failure, and any other condition which, in the opinion of the investigator, would put the subject at risk by participation in the protocol.
6. Hemoglobin <10.0 g/dL, WBC <3.0 x 103/mm3, platelet count <125 x 103/mm3, creatinine > 1.5mg/dL, AST/ALT >2 x ULN, alkaline phosphatase >2 x ULN
7. Known HIV antibody, hepatitis B surface antigen and/or hepatitis C antibody.
8. History of malignancy within 5 years prior to study entry other than carcinoma in situ of the cervix, or adequately treated, non-metastatic squamous or basal cell carcinoma of the skin.
9. History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies.
10. History of tuberculosis (latent or active) or positive Interferon-gamma release assay (IGRA)
11. Infectious disease:

    CRP >30 mg/L, fever, or infection requiring treatment with antibiotics within 3 weeks prior to Screening
12. Immunodeficiency
13. History of treatment with Tysabri or Raptiva
14. Female subjects who are pregnant, planning to become pregnant during the course of the study, or breast-feeding
15. Receipt of a live (attenuated) vaccine within 3 months prior to Screening
16. Major surgery within 28 days prior to Day 0
17. Participation in an investigational drug or device trial within 30 days prior to Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-09-30 (Actual); Primary Completion 2012-07-31 (Actual); Study Completion 2012-08-31 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | 56 days
  Incidence and type of adverse clinical events

SECONDARY OUTCOMES:
RA-18C3 Pharmacokinetics | 56 days
  Serum levels of RA-18C3 will be measured to determine drug half-life, bioavailability, volume of distribution, and area under the curve.
Psoriasis Area and Severity Index (PASI) | 56 days
  Percentage of subjects that acheive PASI 50, PASI 75, and PASI 90
Erythrocyte Sedimentation Rate | 56 days
Physician's Global Assessment Score (PGA) | 56 days
  Change in PGA from baseline to day 56
Dermatology Life Quality Index Questionnaire (DLQI) | 56 days
  Change in DLQI from baseline to day 56
C-reactive protein | 56 days

CONTACTS AND LOCATIONS:
Overall Officials: Johann Gudjonsson, M.D., PhD, Principal Investigator — University of Michigan
Locations (3):
- United States (3):
  - West Kentucky Dermatology, Owensboro, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - Westlake Dermatology, Austin, Texas